CLINICAL TRIAL: NCT00309647
Title: A Partially-blind Multi-centric Study in Adults Aged Between 18-60 Years Designed to Evaluate the Reactogenicity and Immunogenicity of 1 and 2 Doses of Pandemic Monovalent (H5N1) Influenza Vaccines (Whole Virus Formulation) Administered at Different Doses and Adjuvanted or Not
Brief Title: Study to Evaluate the Safety and Immunogenicity of Pandemic Monovalent (H5N1) Influenza Vaccines (Whole Virus Formulation) in Adults 18 and 60 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 106378
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: prophylaxis of pandemic influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (8):
- H5N1 Formulation 1 Group (Experimental): Subjects in this group received 2 doses of H5N1 adjuvanted formulation 1 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1) adjuvanted vaccine
- H5N1 Formulation 2 Group (Experimental): Subjects in this group received 2 doses of H5N1 adjuvanted formulation 2 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1) adjuvanted vaccine
- H5N1 Formulation 3 Group (Experimental): Subjects in this group received 2 doses of H5N1 adjuvanted formulation 3 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1) adjuvanted vaccine
- H5N1 Formulation 4 Group (Experimental): Subjects in this group received 2 doses of H5N1 adjuvanted formulation 4 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1) adjuvanted vaccine
- H5N1 Formulation 5 Group (Active Comparator): Subjects in this group received 2 doses of H5N1 formulation 5 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1)
- H5N1 Formulation 6 Group (Active Comparator): Subjects in this group received 2 doses of H5N1 formulation 6 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1)
- H5N1 Formulation 7 Group (Active Comparator): Subjects in this group received 2 doses of H5N1 formulation 7 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1)
- H5N1 Formulation 8 Group (Active Comparator): Subjects in this group received 2 doses of H5N1 formulation 8 vaccine at a 21-day interval
  Interventions: Biological: Influenza Monovalent Whole virus (H5N1)

INTERVENTIONS:
Biological: Influenza Monovalent Whole virus (H5N1) adjuvanted vaccine — 2 doses administered intramuscularly at the deltoid region of the non-dominant arm at Days 0 and 21
  Arms: H5N1 Formulation 1 Group; H5N1 Formulation 2 Group; H5N1 Formulation 3 Group; H5N1 Formulation 4 Group
Biological: Influenza Monovalent Whole virus (H5N1) — 2 doses administered intramuscularly at the deltoid region of the non-dominant arm at Days 0 and 21
  Arms: H5N1 Formulation 5 Group; H5N1 Formulation 6 Group; H5N1 Formulation 7 Group; H5N1 Formulation 8 Group

SUMMARY:
Today, the leading contender for the next pandemic of influenza is H5N1, a strain of avian virus. Prevention and control of a pandemic will depend on the rapid production and worldwide distribution of specific pandemic vaccines. Candidate 'pandemic-like' vaccines must be developed and tested in clinical trials to determine the most optimal formulation and the best vaccination schedule.This study is designed to test in healthy adults aged between 18-60 years the reactogenicity and immunogenicity of one and two administrations of a candidate pandemic H5N1 vaccine formulated from Whole Virus. The vaccines contain different antigen doses. For each dose, adjuvanted vaccine will be compared to the plain vaccine in order to detect the optimal formulation for immunization against the H5N1 influenza strain.

ELIGIBILITY:
Inclusion criteria:

* A male or female between, and including, 18 and 60 years of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential.

Exclusion criteria:

* Administration of any vaccine during the period starting 15 days before the first administration of the study vaccine and ending 21 after the second one.
* Administration of an influenza vaccine other than the study vaccines during the entire study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or during the study.
* lactating women
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first vaccination, or planned use during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2006-03-29 (Actual); Primary Completion 2006-11-01 (Actual); Study Completion 2006-11-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the humoral immune response induced by the study vaccines in term of anti-haemagglutinin antibody titers | At Days 0, 21, 42 and 180
  Geometric mean titers (GMTs) of serum antibodies
To evaluate the humoral immune response induced by the study vaccines in terms of seroconversion rates (SCRs), Conversion factors and protection rates to H5N1 virus | At days 21, 42 and 180
Occurrence of solicited local and general adverse events | During a 7 day follow-up period (i.e. day of vaccination and 6 subsequent days) after each dose of vaccine and overall
Occurrence of unsolicited adverse events | During a 21 day follow-up period after the first vaccination and 30 day follow-up period after the second vaccination
Occurrence of serious adverse events | During the entire study (Days 0 to 180)

SECONDARY OUTCOMES:
To evaluate the humoral immune response induced by the study vaccines in term of serum neutralizing antibody titers | At Days 0, 21, 42 and 180
  Geometric mean titers (GMTs) of serum antibodies
To evaluate the cell-mediated immune response induced by the study vaccines in term of frequency of influenza-specific CD4/CD8 T lymphocytes | At days 0, 21, 42 and 180
To evaluate the humoral immune response induced by the study vaccines in terms of SCR for serum neutralizing antibody titers | At Days 21, 42 and 180

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Germany (8):
  - GSK Investigational Site, Finsterwalde, Brandenburg
  - GSK Investigational Site, Tostedt, Lower Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Geringswalde, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Elmshorn, Schleswig-Holstein

REFERENCES:
- See also: Results for study 106378 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/106378?search=study&b%22b''%22#rs